CLINICAL TRIAL: NCT06257472
Title: Efficacy of Virtual Reality (VR) for Irritable Bowel Syndrome: A Randomized Trial Comparing Brain-Gut Directed VR vs. Sham VR
Brief Title: Efficacy of Virtual Reality (VR) for Irritable Bowel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborator is taking lead; Entry is now duplicate
Sponsor: Anthony Lembo (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor-Investigator, Anthony Lembo, Vice Chair of Research, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VR Study
Record Dates: First submitted 2024-01-30; First posted 2024-02-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: Virtual Reality; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Two-armed blinded clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS/VR Program (SynerGI) (Experimental)
  Interventions: Device: Virtual Reality Headset
- Sham VR Program (Sham Comparator)
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — Participants will be mailed a Meta Quest 2 Headset. Participants will be asked to wear and use the VR headset for around 20 minutes each day for 8 weeks.

SUMMARY:
In this study, the investigators conduct a remote, eight-week, two-arm, randomized controlled trial that assesses the benefits, primarily measured through the irritable bowel syndrome (IBS)-targeted HRQOL (health-related quality of life), of an immersive, disease-targeted virtual reality program compared to a non-immersive virtual reality program for patients with IBS.

DETAILED DESCRIPTION:
In this study, the investigators will conduct a decentralized, remote, eight-week, two-arm, randomized controlled trial of SynerGI, a disease-targeted, brain-gut directed, immersive VR program for people with IBS, versus sham VR delivered in a VR headset. Eligible participants will be assigned to a study arm using a 1:1 random number generator and will be blinded to allocation. Data analysts will also be blinded to allocation; only pre-specified staff who are uninvolved with data analyses will be unblinded for purposes of study administration (e.g., sending allocation-specific study materials). After completion of the treatment, participants will be invited to participate in an optional 30-minute semi-structured interview to better understand their experiences of VR treatment. Qualitative interviews will be audio-recorded and transcribed.

The primary aim of this study will be to assess the benefits of disease-targeted VR compared to sham VR on clinically relevant outcomes. The second aim will seek to determine patient-level predictors of treatment response to active VR therapy. The third aim will seek to understand patient experiences of VR to better inform the design of VR treatments for digestive diseases in the future.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 18 years or older
* Meet Rome IV criteria, as diagnosed either by a licensed physician or via self-report using the Rome IBS questionnaire, for IBS for any type: IBS-C (IBS with constipation), IBS-D (IBS with diarrhea), and IBS-M (mixed-type IBS)

Exclusion Criteria:

* Individuals with a comorbid disorder that may confound the diagnosis of IBS, including:
* celiac disease
* inflammatory bowel disease
* autoimmune disorders that affect the GI system
* history of bowel resection
* HIV/AIDS ( human immunodeficiency virus/acquired immunodeficiency syndrome)
* diabetes with HgA1c>7.0
* neuroendocrine tumors
* microscopic colitis
* lactase deficiency
* eosinophilic bowel disease
* acute intermittent porphyria
* any other condition that a licensed physician believes can mimic IBS symptoms and undermine diagnostic certitude
* Patients using regular doses of opioid medications will also be excluded given the often-severe impact of opioids on GI motility and potential for pharmacological visceral hyperalgesia
* No WiFi at home
* Any history of seizure
* Ongoing treatment for a GI cancer
* Major audiovisual impairment (complete blindness, deafness)
* Inability to understand English at 6th grade level
* Any events planned over the 8 weeks of the study that could end your ability to participate in the study, such as a medical procedure, vacation, or change in residence (Note: the study team can always delay enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
IBS-targeted HRQOL (health-related quality of life) | Baseline, after 4 weeks using device, after 8 weeks using device
  The primary outcome will be an increase in IBS-QOL (quality of life) scores between baseline and week 8 for those on the study arm. Each question is positively scored 1-5, and the sum is normalized into a 0-100 score, with 100 being the highest reported quality of life and 0 being the lowest.

SECONDARY OUTCOMES:
GI (Gastrointestinal) Pain Intensity | Baseline, after 4 weeks using device, after 8 weeks using device
  A secondary outcome will be a decrease in PROMIS (Patient Reported Outcomes Measurement Information System) GI Pain scores scored on a scale of 1-5 with 1 being low pain intensity and 5 being high. These scores are summed for a raw score, which may be converted into a T-score.
IBS symptom severity | Weekly for 8 weeks
  A secondary outcome will be a decrease in patient reported IBS Symptom Severity Score (IBS-SSS).
  Scored on a 0-500 scale.
  * < 75 points - IBS considered in remission
  * 75-174 - mild IBS
  * 175-299 - moderate IBS
  * 300-500 - severe IBS
    5 measures
    1. # of days with abdominal pain x 10 - maximum score of 100
    2. 1-100 scale for abdominal pain severity
    3. 0-100 scale for abdominal distension severity
    4. 0-100 scale for satisfaction with bowel habits
    5. 0-100 scale for interference with life'
Visceral anxiety | Baseline, after 4 weeks using device, after 8 weeks using device
  A secondary outcome will be a decrease in patient reported Visceral Sensitivity Index (VSI) scores.
  Each question is positively scored 1-6. 1 represents the most visceral anxiety and 6 represents no visceral anxiety.
  The VSI items then are reversed scored, meaning that the 1-6 becomes 5-0. These reverse scores are then summed. The max score, representing severe visceral anxiety is 75. The minimum score is 0 (no visceral anxiety).
Generalized anxiety | Baseline, after 4 weeks using device, after 8 weeks using device
  A secondary outcome will be a decrease in PROMIS (Patient Reported Outcomes Measurement Information System) Anxiety scores. Each question is positively scored 1-5 (meaning that 1 is no anxiety and 5 the highest anxiety), then summed for raw score, which may be converted into a T-Score.
Maladaptive GI (Gastrointestinal) cognitions | Baseline, after 4 weeks using device, after 8 weeks using device
  A secondary outcome will be a decrease in patient reported Gastrointestinal Cognitions Questionnaire (GI-COG) scores.
  Each question is scored positively from 0-4, then summed for raw score. Raw scores 0-19, 20-39, and 40-64 indicate mild catastrophizing, moderate catastrophizing, and severe catastrophizing respectively.
Somatization | Baseline, after 4 weeks using device, after 8 weeks using device
  A secondary outcome will be a decrease in patient reported Patient Health Questionnaire (PHQ-15) scores.
  Each question is positively scored 0-2, then summed for raw score. The total PHQ-15 score ranges from 0 to 30 and scores of ≥5, ≥10, ≥15 represent mild, moderate and severe levels of somatization, respectively.
Increase in Symptom Relief | End of Study, which will occur after 8 weeks using device
  A secondary outcome will be an increase in patient reported "Adequate Relief" global assessment. This is a binary outcome (yes or no)
Optional Individual Cognitive Interviews | End of Study, which will occur after 8 weeks using device
  Obtaining qualitative feedback from participants in the treatment group about their experiences with the SynerGI software
Optional Rome IV Criteria assessment | At screening/baseline
  Using the fourth version of the Rome Criteria, potential participants may self-diagnose themselves with IBS.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cleveland Clinic Main Campus, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No